CLINICAL TRIAL: NCT05496231
Title: A Phase 1/2 Randomized, Observer-blinded, Multi-country Study to Evaluate Safety and Immunogenicity of Investigational Adjuvanted Human Papillomavirus Vaccine in Females (16 to 26 Years of Age)
Brief Title: A Study on the Immune Response and Safety of an Adjuvanted Human Papillomavirus Vaccine When Given to Healthy Women 16 to 26 Years of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 213749; 2022-000090-15 (EudraCT Number)
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Human papillomavirus; Infection; Vaccine; Women's health
MeSH Terms: conditions — Uterine Cervical Dysplasia; Infections | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blinded for study vs comparator vaccine; double-blinded for 3 formulations of study vaccine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- HPV9 High Group (Experimental): Participants received 3 doses of the high formulation of Human Papilloma Virus 9-valent (HPV9) investigational adjuvanted vaccine at Day 1, Month 2, and Month 6.
  Interventions: Biological: HPV9 High formulation
- HPV9 Med Group (Experimental): Participants received 3 doses of the medium formulation of Human Papilloma Virus 9-valent (HPV9) investigational adjuvanted vaccine at Day 1, Month 2, and Month 6.
  Interventions: Biological: HPV9 Medium formulation
- HPV9 Low Group (Experimental): Participants received 3 doses of the low formulation of Human Papilloma Virus 9-valent (HPV9) investigational adjuvanted vaccine at Day 1, Month 2, and Month 6.
  Interventions: Biological: HPV9 Low formulation
- Gar9 Group (Active Comparator): Participants received 3 doses of the marketed Human Papilloma Virus (HPV) vaccine (Gardasil 9) at Day 1, Month 2, and Month 6.
  Interventions: Biological: Gardasil 9

INTERVENTIONS:
Biological: HPV9 High formulation — 3 doses of the high formulation of HPV9 investigational adjuvanted vaccine were administered intramuscularly at Day 1, Month 2 and Month 6.
  Arms: HPV9 High Group
Biological: HPV9 Medium formulation — 3 doses of the medium formulation of HPV9 investigational adjuvanted vaccine were administered intramuscularly at Day 1, Month 2 and Month 6.
  Arms: HPV9 Med Group
Biological: HPV9 Low formulation — 3 doses of the low formulation of HPV9 investigational adjuvanted vaccine were administered intramuscularly at Day 1, Month 2 and Month 6.
  Arms: HPV9 Low Group
Biological: Gardasil 9 — 3 doses of the marketed HPV vaccine (Gardasil 9) were administered intramuscularly at Day 1, Month 2 and Month 6.
  Arms: Gar9 Group

SUMMARY:
The main purpose of this study was to evaluate the safety and reactogenicity of GlaxoSmithKline Biologicals SA (GSK)'s investigational adjuvanted human papillomavirus (HPV) vaccine formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants as established by medical history and clinical examination before entering into the study.
2. For Step 1 only: Female between and including 18 and 26 years of age at the time of the first study intervention administration.
3. For Step 2: Female between and including 16 and 26 years of age at the time of the first study intervention administration.
4. Written informed consent obtained from the participant prior to performance of any study specific procedure (for participants below the legal age of consent as per local regulations, written informed consent must be obtained from the participant/participant's parent[s]/legally authorized representatives [LAR{s}] and, in addition, the participant should sign and personally date a written informed assent).
5. Participants and/or participants' parent(s)/LAR(s) who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiary, return for follow-up visits).
6. Female participant with no more than 4 lifetime sexual partners prior to enrollment.
7. Female participants of non-childbearing potential may be enrolled in the study.

Female participants of childbearing potential may be enrolled in the study if the participant:

* has practiced adequate highly effective contraception for at least 1 month prior to study intervention administration, and
* has a negative pregnancy test on the day of study intervention administration, and
* has agreed to continue adequate contraception during the entire intervention period and for 2 months after completion of the study intervention administration series.

Exclusion Criteria:

1. Pregnant or lactating female.
2. Female planning to become pregnant or planning to discontinue contraceptive precautions.
3. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
4. History or current diagnosis of autoimmune disease.
5. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
6. Hypersensitivity to latex.
7. Major congenital defects, as assessed by the investigator.
8. History of abnormal Papanicolaou test or abnormal cervical biopsy result.
9. History of external genital/vaginal warts.
10. History of positive HPV test.
11. Acute or chronic clinically significant pulmonary, cardiovascular, neurologic, hepatic or renal functional abnormality, as determined by physical examination or laboratory tests
12. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
13. Previous vaccination against HPV.
14. Previous exposure to monophosphoryl lipid A (MPL) or AS04 adjuvant.
15. Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study intervention(s) during the period beginning 30 days before the first dose of study intervention(s) (Day -29 to Day 1), or their planned use during the study period.
16. Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before each dose and ending 30 days after each dose of study interventions administration*

    *In case emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is organized by public health authorities outside the routine immunization program, the time period described above can be reduced if, necessary for that vaccine, provided it is licensed and used according to its Product Information.
17. Administration of long-acting immune-modifying drugs at any time during the study period.
18. Use of systemic cytotoxic agents within the previous 3 months prior to randomization into this study or at any time during the study period.
19. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first study intervention dose(s). For corticosteroids, this will mean prednisone equivalent ≥20 mg/day for adult participants/ ≥0.5 milligram/kilogram/day (mg/kg/day) with maximum of 20 mg/day for participants under 18 years of age. Inhaled and topical steroids are allowed.
20. Administration of systemic immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the administration of the first dose of study interventions or planned administration during the study period.
21. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non investigational intervention.
22. History of /current chronic alcohol consumption and/or drug abuse.
23. Any study personnel or their immediate dependents, family, or household members.
24. Child in care.

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only female participants, between 16-26 years of age were included in the study.
Enrollment: 1080 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (36):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami Beach, Florida
  - GSK Investigational Site, Pompano Beach, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Saginaw, Michigan
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Norman, Oklahoma
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Carrollton, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Humble, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Norfolk, Virginia
- GSK Investigational Site, Sofia, Bulgaria
- Czechia (3):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (7):
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, La Roche-sur-Yon
  - GSK Investigational Site, La Tronche
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Tours
- Germany (2):
  - GSK Investigational Site, Schwerin
  - GSK Investigational Site, Würzburg
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was organized into 2 steps. Step 1 sentinel participants received the initial assigned dose prior to participants in Step 2 of the study, and sentinel participants had an additional blood sampling visit at Day 7 to assess for biochemical and hematological parameters.
Pre-assignment Details: A total of 1080 participants were enrolled into the study, of which 1079 participants received at least 1 dose of vaccine and were included in the Exposed Set.
Period: Overall Study
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Started | 270 | 270 | 269 | 270
Completed | 239 | 246 | 244 | 238
Not Completed | 31 | 24 | 25 | 32
Not completed — Adverse Event | 1 | 1 | 0 | 4
Not completed — Withdrawal by Subject | 5 | 5 | 4 | 11
Not completed — Migrated/moved from the study area | 3 | 5 | 3 | 3
Not completed — Lost to Follow-up | 13 | 6 | 11 | 6
Not completed — Other | 9 | 7 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group | Total
Number analyzed (Participants) | 270 | 270 | 269 | 270 | 1079
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.0 (2.32) | 21.9 (2.56) | 22.1 (2.45) | 22.2 (2.25) | 22.1 (2.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 270 | 270 | 269 | 270 | 1079
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 25 | 27 | 26 | 103
  Not Hispanic or Latino | 245 | 245 | 242 | 244 | 976
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Grade 3 Solicited Administration Site Events After Vaccine Dose 1
Description: Assessed solicited administration site events included pain, redness and swelling at injection site. Grade 3 pain = significant pain at rest, which prevented normal everyday activities. Grade 3 redness/swelling = redness/swelling with a surface diameter greater than (>) 50 millimeters (mm).
Time Frame: Within 7 days after vaccine Dose 1 (administered at Day 1)
Population: Analysis was performed on the Exposed Set, which included all participants who received a study vaccine, had the electronic diary (eDiary) for solicited events completed after the administration of vaccine Dose 1 and for whom data were available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 270 | 270 | 269 | 270
Participants
  Grade 3 Pain | 11 | 12 | 6 | 2
  Grade 3 Redness | 2 | 4 | 2 | 0
  Grade 3 Swelling | 5 | 3 | 2 | 0

2. Primary Outcome: Number of Participants Reporting Grade 3 Solicited Administration Site Events After Vaccine Dose 2
Description: Assessed solicited administration site events included pain, redness and swelling at injection site. Grade 3 pain = significant pain at rest, which prevented normal everyday activities. Grade 3 redness/swelling = redness/swelling with a surface diameter >50 mm.
Time Frame: Within 7 days after vaccine Dose 2 (administered at Month 2)
Population: Analysis was performed on the Exposed Set, which included all participants who received a study vaccine, had the eDiary for solicited events completed after the administration of vaccine Dose 2 and for whom data were available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 257 | 261 | 258 | 260
Participants
  Grade 3 Pain | 13 | 6 | 11 | 1
  Grade 3 Redness | 4 | 0 | 2 | 1
  Grade 3 Swelling | 5 | 3 | 2 | 3

3. Primary Outcome: Number of Participants Reporting Grade 3 Solicited Administration Site Events After Vaccine Dose 3
Description: as for outcome 2
Time Frame: Within 7 days after vaccine Dose 3 (administered at Month 6)
Population: Analysis was performed on the Exposed Set, which included all participants who received a study vaccine, had the eDiary for solicited events completed after the administration of vaccine Dose 3 and for whom data were available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 244 | 247 | 244 | 236
Participants
  Grade 3 Pain | 9 | 3 | 6 | 1
  Grade 3 Redness | 0 | 2 | 1 | 1
  Grade 3 Swelling | 0 | 4 | 1 | 2

4. Primary Outcome: Number of Participants Reporting Grade 3 Solicited Systemic Events After Vaccine Dose 1
Description: Assessed solicited systemic events included fever, headache, myalgia, arthralgia and fatigue. Grade 3 fever = body temperature >39.0 degrees Celsius (°C) or 102.2 Fahrenheit (°F). The preferred location for measuring temperature was the axilla. Grade 3 headache, myalgia, arthralgia and fatigue = symptoms that prevented normal, every day activities.
Time Frame: Within 7 days after vaccine Dose 1 (administered at Day 1)
Population: Analysis was performed on the Exposed Set, which included all participants who received a study vaccine, had the eDiary for solicited events completed after the administration of vaccine Dose 1 and for whom data were available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 270 | 270 | 269 | 270
Participants
  Grade 3 Fever | 1 | 0 | 0 | 0
  Grade 3 Headache | 11 | 3 | 6 | 3
  Grade 3 Myalgia | 5 | 2 | 2 | 1
  Grade 3 Arthralgia | 1 | 1 | 1 | 0
  Grade 3 Fatigue | 12 | 9 | 7 | 5

5. Primary Outcome: Number of Participants Reporting Grade 3 Solicited Systemic Events After Vaccine Dose 2
Description: Assessed solicited systemic events included fever, headache, myalgia, arthralgia and fatigue. Grade 3 fever = body temperature >39.0°C or 102.2°F. The preferred location for measuring temperature was the axilla. Grade 3 headache, myalgia, arthralgia and fatigue = symptoms that prevented normal, every day activity.
Time Frame: Within 7 days after vaccine Dose 2 (administered at Month 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 257 | 261 | 258 | 260
Participants
  Grade 3 Fever | 0 | 1 | 0 | 1
  Grade 3 Headache | 7 | 7 | 8 | 5
  Grade 3 Myalgia | 4 | 0 | 3 | 2
  Grade 3 Arthralgia | 0 | 2 | 1 | 1
  Grade 3 Fatigue | 12 | 11 | 12 | 11

6. Primary Outcome: Number of Participants Reporting Grade 3 Solicited Systemic Events After Vaccine Dose 3
Description: as for outcome 5
Time Frame: Within 7 days after vaccine Dose 3 (administered at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 244 | 247 | 244 | 236
Participants
  Grade 3 Fever | 0 | 1 | 0 | 0
  Grade 3 Headache | 10 | 4 | 9 | 7
  Grade 3 Myalgia | 3 | 3 | 2 | 2
  Grade 3 Arthralgia | 2 | 1 | 0 | 0
  Grade 3 Fatigue | 15 | 8 | 11 | 6

7. Primary Outcome: Number of Participants Reporting Grade 3 Unsolicited Adverse Events (AEs) After Vaccine Dose 1
Description: An unsolicited AE is defined as an AE that was not included in the list of solicited events using an eDiary and that was spontaneously communicated by a participant/participant's parent(s)/legally acceptable representative(s) [LAR(s)] who has signed the informed consent. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE. Grade 3 unsolicited AEs = an AE which prevented normal, everyday activities.
Time Frame: Within 28 days after vaccine Dose 1 (administered at Day 1)
Population: Analysis was performed on the Exposed Set, which included all participants who received a study vaccine and for whom data were available for the specified period after the administration of vaccine Dose 1.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 270 | 270 | 269 | 270
Participants | 0 | 1 | 0 | 1

8. Primary Outcome: Number of Participants Reporting Grade 3 Unsolicited AEs After Vaccine Dose 2
Description: An unsolicited AE is defined as an AE that was not included in the list of solicited events using an eDiary and that was spontaneously communicated by a participant/participant's parent(s)/LAR(s) who has signed the informed consent. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE. Grade 3 unsolicited AEs = an AE which prevented normal, everyday activities.
Time Frame: Within 28 days after vaccine Dose 2 (administered at Month 2)
Population: Analysis was performed on the Exposed Set, which included all participants who received a study vaccine and for whom data were available for the specified period after the administration of vaccine Dose 2.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 257 | 261 | 258 | 260
Participants | 4 | 1 | 3 | 3

9. Primary Outcome: Number of Participants Reporting Grade 3 Unsolicited AEs After Vaccine Dose 3
Description: An unsolicited AE is defined as an AE that was not included in the list of solicited events using an eDiary and that was spontaneously communicated by a participant/ participant's parent(s)/LAR(s) who has signed the informed consent. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE. Grade 3 unsolicited AEs = an AE which prevented normal, everyday activities.
Time Frame: Within 28 days after vaccine Dose 3 (administered at Month 6)
Population: Analysis was performed on the Exposed Set, which included all participants who received a study vaccine and for whom data were available for the specified period after the administration of vaccine Dose 3.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 244 | 247 | 244 | 236
Participants | 0 | 0 | 1 | 2

10. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant, or resulted in abnormal pregnancy outcomes, or in other situations that were considered serious per medical or scientific judgment.
Time Frame: From first vaccination (Day 1) to study end (Month 12)
Population: Analysis was performed on the Exposed Set, which included participants who received a study vaccine and for whom data were available for the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 270 | 270 | 269 | 270
Participants | 1 | 4 | 2 | 7

11. Primary Outcome: Number of Participants in Step 1 Subset With Clinically Relevant Biochemical Abnormalities
Description: As pre-specified in the protocol, the assessed biochemical parameters were blood urea nitrogen (BUN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST). Assessment of intensity: Grading of the biochemical parameters was based on the institutional normal reference ranges and derived from the standard Food and Drug Administration (FDA) Toxicity Grading Scale. Changes compared to normal reference ranges were graded as follows: Grade 0 = a non-missing parameter value for which grade could not be derived according to the grading scale and does not belong to Grade 1-4; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life-Threatening. Unknown = parameter value missing for the specified parameter.
Time Frame: At Day 7
Population: Analysis was performed on the Step 1 subset from the Exposed Set, which included sentinel adult participants for whom blood samples were collected for the specified biochemical analyses at Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  BUN, Grade 0 | 11 | 12 | 11 | 11
  BUN, Grade 1 | 0 | 0 | 0 | 0
  BUN, Grade 2 | 0 | 0 | 0 | 0
  BUN, Grade 3 | 0 | 0 | 0 | 0
  BUN, Grade 4 | 0 | 0 | 0 | 0
  BUN, Unknown | 1 | 0 | 1 | 1
  AST, Grade 0 | 11 | 12 | 11 | 12
  AST, Grade 1 | 0 | 0 | 0 | 0
  AST, Grade 2 | 0 | 0 | 0 | 0
  AST, Grade 3 | 0 | 0 | 0 | 0
  AST, Grade 4 | 0 | 0 | 0 | 0
  AST, Unknown | 1 | 0 | 1 | 0
  ALT, Grade 0 | 11 | 12 | 11 | 12
  ALT, Grade 1 | 0 | 0 | 0 | 0
  ALT, Grade 2 | 0 | 0 | 0 | 0
  ALT, Grade 3 | 0 | 0 | 0 | 0
  ALT, Grade 4 | 0 | 0 | 0 | 0
  ALT, Unknown | 1 | 0 | 1 | 0

12. Primary Outcome: Number of Participants in Step 1 Subset With Clinically Relevant Hematological Abnormalities
Description: As pre-specified in the protocol, the assessed hematological parameters were hemoglobin, white blood cells (WBC) increase, WBC decrease, lymphocyte decrease, neutrophils decrease, eosinophils, and platelets decrease. Assessment of intensity: Grading of the biochemical parameters was based on the institutional normal reference ranges and derived from the standard FDA Toxicity Grading Scale. Changes compared to normal reference ranges were graded as follows: Grade 0 = a non-missing parameter value for which grade could not be derived according to the grading scale and does not belong to Grade 1-4; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life-Threatening; Unknown = parameter value missing for the specified parameter.
Time Frame: At Day 7
Population: Analysis was performed on the Step 1 subset from the Exposed Set, which included sentinel adult participants for whom blood samples were collected for the specified hematological analyses at Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Hemoglobin, Grade 0 | 8 | 10 | 9 | 8
  Hemoglobin, Grade 1 | 3 | 1 | 2 | 4
  Hemoglobin, Grade 2 | 0 | 0 | 0 | 0
  Hemoglobin, Grade 3 | 0 | 1 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin, Unknown | 1 | 0 | 1 | 0
  WBC Increase, Grade 0 | 11 | 12 | 11 | 11
  WBC Increase, Grade 1 | 0 | 0 | 0 | 1
  WBC Increase, Grade 2 | 0 | 0 | 0 | 0
  WBC Increase, Grade 3 | 0 | 0 | 0 | 0
  WBC Increase, Grade 4 | 0 | 0 | 0 | 0
  WBC Increase, Unknown | 1 | 0 | 1 | 0
  WBC Decrease, Grade 0 | 11 | 11 | 10 | 11
  WBC Decrease, Grade 1 | 0 | 1 | 1 | 1
  WBC Decrease, Grade 2 | 0 | 0 | 0 | 0
  WBC Decrease, Grade 3 | 0 | 0 | 0 | 0
  WBC Decrease, Grade 4 | 0 | 0 | 0 | 0
  WBC Decrease, Unknown | 1 | 0 | 1 | 0
  Lymphocyte Decrease, Grade 0 | 11 | 12 | 11 | 12
  Lymphocyte Decrease, Grade 1 | 0 | 0 | 0 | 0
  Lymphocyte Decrease, Grade 2 | 0 | 0 | 0 | 0
  Lymphocyte Decrease, Grade 3 | 0 | 0 | 0 | 0
  Lymphocyte Decrease, Grade 4 | 0 | 0 | 0 | 0
  Lymphocyte Decrease, Unknown | 1 | 0 | 1 | 0
  Neutrophils Decrease, Grade 0 | 10 | 11 | 10 | 11
  Neutrophils Decrease, Grade 1 | 1 | 0 | 1 | 1
  Neutrophils Decrease, Grade 2 | 0 | 1 | 0 | 0
  Neutrophils Decrease, Grade 3 | 0 | 0 | 0 | 0
  Neutrophils Decrease, Grade 4 | 0 | 0 | 0 | 0
  Neutrophils Decrease, Unknown | 1 | 0 | 1 | 0
  Eosinophils, Grade 0 | 11 | 12 | 11 | 11
  Eosinophils, Grade 1 | 0 | 0 | 0 | 1
  Eosinophils, Grade 2 | 0 | 0 | 0 | 0
  Eosinophils, Grade 3 | 0 | 0 | 0 | 0
  Eosinophils, Grade 4 | 0 | 0 | 0 | 0
  Eosinophils, Unknown | 1 | 0 | 1 | 0
  Platelet Decrease, Grade 0 | 11 | 12 | 11 | 12
  Platelet Decrease, Grade 1 | 0 | 0 | 0 | 0
  Platelet Decrease, Grade 2 | 0 | 0 | 0 | 0
  Platelet Decrease, Grade 3 | 0 | 0 | 0 | 0
  Platelet Decrease, Grade 4 | 0 | 0 | 0 | 0
  Platelet Decrease, Unknown | 1 | 0 | 1 | 0

13. Primary Outcome: Number of Participants in Step 1 Subset With Clinically Relevant Abnormalities in Hemoglobin Change From Baseline Levels
Description: The number of participants with clinically relevant abnormalities in hemoglobin change from baseline levels is reported. Assessment of intensity: Grading of the biochemical parameters was based on the institutional normal reference ranges and derived from the standard FDA Toxicity Grading Scale. Changes compared to normal reference ranges were graded as follows: Grade 0 = a non-missing parameter value for which grade could not be derived according to the grading scale and does not belong to Grade 1-4; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life-Threatening; Unknown = parameter value missing for the specified parameter. Change from baseline = the difference between a participant's baseline (pre-intervention) parameter values and their follow-up (post-intervention) parameter values.
Time Frame: At Day 7 compared to baseline (Day 1)
Population: Analysis was performed on the Step 1 subset from the Exposed Set, which included sentinel adult participants for whom blood samples were collected for the hemoglobin change from baseline analysis at Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Hemoglobin change from baseline, Grade 0 | 5 | 1 | 1 | 5
  Hemoglobin change from baseline, Grade 1 | 5 | 11 | 8 | 6
  Hemoglobin change from baseline, Grade 2 | 0 | 0 | 1 | 0
  Hemoglobin change from baseline, Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin change from baseline, Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin change from baseline, Unknown | 2 | 0 | 2 | 1

14. Primary Outcome: Anti-HPV Immunoglobulin G (IgG) Antibody Concentrations
Description: Anti-HPV IgG antibody concentrations were determined by electrochemiluminescence (ECL) assay and expressed as geometric mean concentrations (GMCs) in arbitrary units per milliliter (AU/mL). The assessed antigens were: HPV 6, HPV 11, HPV 16, HPV 18, HPV 31, HPV 33, HPV 45, HPV 52 and HPV 58 type antigens.
Time Frame: At Month 7 (one month after vaccine Dose 3 administration)
Population: Analysis was performed on Per Protocol Set (PPS) for immunogenicity, which included all participants from Exposed Set who met all eligibility criteria, followed the protocol for vaccine administration, adhered to vaccination schedule and blood sampling timings, and had post-vaccination immunogenicity results available for the specified analysis at the specified time point. The PPS excluded those participants with protocol deviations, interfering medications, or intercurrent medical conditions.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 211 | 201 | 206 | 203
AU/mL
  HPV 6 type antigen: number analyzed (Participants) | 210 | 201 | 206 | 203
  HPV 6 type antigen | 124141.35 [110854.94 to 139020.20] | 117881.81 [103701.90 to 134000.65] | 119724.25 [105236.23 to 136206.84] | 54710.66 [47259.35 to 63336.80]
  HPV 11 type antigen: number analyzed (Participants) | 211 | 201 | 205 | 203
  HPV 11 type antigen | 276225.68 [243524.62 to 313317.91] | 250405.46 [217218.09 to 288663.30] | 260309.15 [223319.56 to 303425.52] | 187507.09 [162968.13 to 215740.99]
  HPV 16 type antigen: number analyzed (Participants) | 202 | 191 | 202 | 197
  HPV 16 type antigen | 297480.37 [254936.96 to 347123.34] | 272728.60 [231905.67 to 320737.69] | 294326.70 [252346.28 to 343290.99] | 154844.90 [131166.44 to 182797.86]
  HPV 18 type antigen: number analyzed (Participants) | 211 | 200 | 205 | 203
  HPV 18 type antigen | 181939.71 [157766.95 to 209816.17] | 172862.73 [148117.04 to 201742.65] | 183180.47 [156207.11 to 214811.50] | 86756.51 [73744.88 to 102063.92]
  HPV 31 type antigen: number analyzed (Participants) | 211 | 200 | 206 | 203
  HPV 31 type antigen | 241644.97 [215104.30 to 271460.37] | 221590.60 [192869.71 to 254588.41] | 230875.63 [202104.78 to 263742.19] | 104667.37 [90853.53 to 120581.53]
  HPV 33 type antigen: number analyzed (Participants) | 208 | 200 | 198 | 198
  HPV 33 type antigen | 154537.14 [133354.03 to 179085.17] | 146931.12 [125717.81 to 171723.90] | 150919.88 [128301.37 to 177525.85] | 96875.65 [84426.91 to 111159.96]
  HPV 45 type antigen | 170959.55 [149389.05 to 195644.64] | 174740.31 [151200.15 to 201945.41] | 174014.45 [150322.39 to 201440.58] | 71768.92 [61224.65 to 84129.14]
  HPV 52 type antigen: number analyzed (Participants) | 211 | 200 | 206 | 201
  HPV 52 type antigen | 203994.24 [180491.88 to 230556.91] | 196454.98 [172561.35 to 223657.02] | 204005.75 [178367.04 to 233329.81] | 103497.80 [90571.68 to 118268.69]
  HPV 58 type antigen: number analyzed (Participants) | 210 | 199 | 205 | 202
  HPV 58 type antigen | 193735.34 [167223.71 to 224450.13] | 186513.90 [161169.95 to 215843.18] | 190767.16 [162753.08 to 223603.20] | 93456.26 [80147.35 to 108975.18]

15. Secondary Outcome: Number of Participants Reporting Any Solicited Administration Site Events
Description: Assessed solicited administration site events included pain, redness and swelling at injection site. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: Within 7 days after each vaccine dose (administered at Day 1, Month 2, and Month 6)
Population: Analysis was performed on the Exposed Set, which included all participants who received a study vaccine, had the eDiary for solicited events completed after the administration of each vaccine dose and for whom data were available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 270 | 270 | 269 | 270
Participants
  Any pain, post-dose 1 | 240 | 244 | 245 | 188
  Any redness, post-dose 1 | 71 | 70 | 91 | 47
  Any swelling, post-dose 1 | 61 | 54 | 66 | 21
  Any pain, post-dose 2: number analyzed (Participants) | 257 | 261 | 258 | 260
  Any pain, post-dose 2 | 208 | 221 | 218 | 185
  Any redness, post-dose 2: number analyzed (Participants) | 257 | 261 | 258 | 260
  Any redness, post-dose 2 | 79 | 83 | 69 | 46
  Any swelling, post-dose 2: number analyzed (Participants) | 257 | 261 | 258 | 260
  Any swelling, post-dose 2 | 68 | 55 | 59 | 35
  Any pain, post-dose 3: number analyzed (Participants) | 244 | 247 | 244 | 236
  Any pain, post-dose 3 | 188 | 191 | 191 | 155
  Any redness, post-dose 3: number analyzed (Participants) | 244 | 247 | 244 | 236
  Any redness, post-dose 3 | 61 | 64 | 64 | 37
  Any swelling, post-dose 3: number analyzed (Participants) | 244 | 247 | 244 | 236
  Any swelling, post-dose 3 | 59 | 52 | 58 | 24

16. Secondary Outcome: Number of Participants Reporting Any Solicited Systemic Events
Description: Assessed solicited systemic events included fever (defined as body temperature >=37.5°C/99.5°F), headache, myalgia, arthralgia and fatigue. The preferred location for measuring temperature was the axilla. Any = occurrence of the symptom regardless of intensity grade or relation to study vaccination.
Time Frame: Within 7 days after each vaccine dose (administered at Day 1, Month 2, and Month 6)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 270 | 270 | 269 | 270
Participants
  Any fever, post-dose 1 | 15 | 12 | 10 | 13
  Any headache, post-dose 1 | 137 | 113 | 131 | 127
  Any myalgia, post-dose 1 | 87 | 105 | 92 | 75
  Any arthralgia, post-dose 1 | 27 | 25 | 22 | 23
  Any fatigue, post-dose 1 | 180 | 166 | 146 | 149
  Any fever, post-dose 2: number analyzed (Participants) | 257 | 261 | 258 | 260
  Any fever, post-dose 2 | 8 | 13 | 9 | 16
  Any headache, post-dose 2: number analyzed (Participants) | 257 | 261 | 258 | 260
  Any headache, post-dose 2 | 113 | 106 | 118 | 101
  Any myalgia, post-dose 2: number analyzed (Participants) | 257 | 261 | 258 | 260
  Any myalgia, post-dose 2 | 80 | 67 | 66 | 56
  Any arthralgia, post-dose 2: number analyzed (Participants) | 257 | 261 | 258 | 260
  Any arthralgia, post-dose 2 | 25 | 19 | 21 | 20
  Any fatigue, post-dose 2: number analyzed (Participants) | 257 | 261 | 258 | 260
  Any fatigue, post-dose 2 | 152 | 132 | 124 | 127
  Any fever, post-dose 3: number analyzed (Participants) | 244 | 247 | 244 | 236
  Any fever, post-dose 3 | 13 | 11 | 11 | 8
  Any headache, post-dose 3: number analyzed (Participants) | 244 | 247 | 244 | 236
  Any headache, post-dose 3 | 106 | 81 | 84 | 85
  Any myalgia, post-dose 3: number analyzed (Participants) | 244 | 247 | 244 | 236
  Any myalgia, post-dose 3 | 61 | 59 | 54 | 45
  Any arthralgia, post-dose 3: number analyzed (Participants) | 244 | 247 | 244 | 236
  Any arthralgia, post-dose 3 | 21 | 15 | 19 | 10
  Any fatigue, post-dose 3: number analyzed (Participants) | 244 | 247 | 244 | 236
  Any fatigue, post-dose 3 | 122 | 103 | 103 | 102

17. Secondary Outcome: Number of Participants Reporting Any Unsolicited AEs
Description: An unsolicited AE is defined as an AE that was not included in the list of solicited events using an eDiary and that was spontaneously communicated by a participant/participant's parent(s)/LAR(s) who has signed the informed consent. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE. Any = occurrence of the symptom regardless of intensity grade or relation to study vaccination.
Time Frame: Within 28 days after each vaccine dose (administered at Day 1, Month 2, and Month 6)
Population: Analysis was performed on the Exposed Set, which included all participants who received a study vaccine and for whom data were available for the specified period after the administration of each vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 270 | 270 | 269 | 270
Participants
  Any unsolicited AEs, post-dose 1 | 70 | 72 | 70 | 70
  Any unsolicited AEs, post-dose 2: number analyzed (Participants) | 257 | 261 | 258 | 260
  Any unsolicited AEs, post-dose 2 | 51 | 38 | 58 | 55
  Any unsolicited AEs, post-dose 3: number analyzed (Participants) | 244 | 247 | 244 | 236
  Any unsolicited AEs, post-dose 3 | 37 | 41 | 45 | 31

18. Secondary Outcome: Number of Participants Reporting Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are defined as a subset of AEs of special interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From first vaccination (Day 1) to study end (Month 12)
Population: Analysis was performed on the Exposed set, which included all participants who received a study vaccine and for whom data were available for the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 270 | 270 | 269 | 270
Participants | 0 | 0 | 2 | 2

19. Secondary Outcome: Number of Participants Reporting Pregnancies
Description: The number of participants who experienced pregnancy while participating in this study is reported.
Time Frame: From Day 1 of pregnancy to study end (Month 12)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 270 | 270 | 269 | 270
Participants | 1 | 3 | 0 | 5

20. Secondary Outcome: Number of Participants With Outcomes of Reported Pregnancies
Description: The participants with confirmed pregnancies were followed up to determine the outcomes of the reported pregnancies. Pregnancy outcomes were live infant, no apparent congenital anomaly; elective termination, no apparent congenital anomaly, and ectopic pregnancy.
Time Frame: From Day 1 of pregnancy up to study end (Month 12)
Population: Analysis was performed on the Exposed set, which included all participants who received a study vaccine, who reported any pregnancy and for whom data were available for the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 1 | 3 | 0 | 5
Participants
  Live infant, no apparent congenital anomaly | 1 | 2 | 0 | 2
  Elective termination, no apparent congenital anomaly | 0 | 1 | 0 | 2
  Ectopic pregnancy | 0 | 0 | 0 | 1

21. Secondary Outcome: Anti-HPV IgG Antibody Concentrations
Description: Anti-HPV IgG antibody concentrations were determined by ECL assay and expressed as GMCs in AU/mL. The assessed antigens were: HPV 6, HPV 11, HPV 16, HPV 18, HPV 31, HPV 33, HPV 45, HPV 52 and HPV 58 type antigens.
Time Frame: At Day 1, Month 2, Month 3, Month 6, Month 7 (Month 7 data was also reported in primary outcome measure 14, as pre-specified in protocol) and Month 12
Population: Analysis was performed on Per Protocol Set (PPS) for immunogenicity, which included all participants from Exposed Set who met all eligibility criteria, followed the protocol for vaccine administration, adhered to vaccination schedule and blood sampling timings, and had post-vaccination immunogenicity results available for the specified analysis at the specified time points. The PPS excluded those participants with protocol deviations, interfering medications, or intercurrent medical conditions.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 265 | 261 | 264 | 261
AU/mL
  HPV 6 type antigen, Day 1: number analyzed (Participants) | 264 | 261 | 263 | 261
  HPV 6 type antigen, Day 1 | 3621.58 [3245.94 to 4040.70] | 3377.84 [3078.74 to 3705.98] | 3124.40 [2891.32 to 3376.27] | 2970.65 [2773.07 to 3182.30]
  HPV 6 type antigen, Month 2: number analyzed (Participants) | 235 | 235 | 234 | 235
  HPV 6 type antigen, Month 2 | 29701.14 [25289.04 to 34883.02] | 29699.92 [25343.87 to 34804.68] | 23870.12 [20301.64 to 28065.86] | 10488.57 [8707.08 to 12634.56]
  HPV 6 type antigen, Month 3: number analyzed (Participants) | 223 | 232 | 231 | 229
  HPV 6 type antigen, Month 3 | 113669.75 [101762.75 to 126969.97] | 106471.07 [95221.75 to 119049.37] | 100258.49 [88766.41 to 113238.38] | 63245.70 [55720.23 to 71787.54]
  HPV 6 type antigen, Month 6: number analyzed (Participants) | 225 | 222 | 220 | 212
  HPV 6 type antigen, Month 6 | 42722.37 [37809.13 to 48274.08] | 38982.11 [34388.98 to 44188.73] | 32792.55 [28876.62 to 37239.51] | 18744.02 [15944.74 to 22034.74]
  HPV 6 type antigen, Month 7: number analyzed (Participants) | 210 | 201 | 206 | 203
  HPV 6 type antigen, Month 7 | 124141.35 [110854.94 to 139020.20] | 117881.81 [103701.90 to 134000.65] | 119724.25 [105236.23 to 136206.84] | 54710.66 [47259.35 to 63336.80]
  HPV 6 type antigen, Month 12: number analyzed (Participants) | 198 | 200 | 197 | 196
  HPV 6 type antigen, Month 12 | 68118.04 [60118.11 to 77182.53] | 65112.37 [56605.42 to 74897.80] | 59776.32 [51986.07 to 68733.97] | 26890.23 [22982.31 to 31462.65]
  HPV 11 type antigen, Day 1: number analyzed (Participants) | 265 | 261 | 263 | 261
  HPV 11 type antigen, Day 1 | 2217.95 [1860.09 to 2644.67] | 2105.07 [1797.78 to 2464.89] | 2013.18 [1725.27 to 2349.12] | 1794.54 [1572.94 to 2047.37]
  HPV 11 type antigen, Month 2: number analyzed (Participants) | 236 | 235 | 230 | 234
  HPV 11 type antigen, Month 2 | 41618.25 [35124.62 to 49312.39] | 37945.17 [32187.34 to 44732.98] | 29437.94 [24557.93 to 35287.68] | 38760.82 [32890.19 to 45679.30]
  HPV 11 type antigen, Month 3: number analyzed (Participants) | 224 | 232 | 230 | 229
  HPV 11 type antigen, Month 3 | 231064.29 [203232.17 to 262707.95] | 212805.15 [185957.86 to 243528.46] | 192296.18 [167234.40 to 221113.72] | 220402.45 [196291.74 to 247474.71]
  HPV 11 type antigen, Month 6: number analyzed (Participants) | 226 | 222 | 219 | 212
  HPV 11 type antigen, Month 6 | 77600.50 [68286.55 to 88184.84] | 67299.61 [58975.99 to 76798.00] | 57076.00 [49315.68 to 66057.49] | 68934.35 [59315.95 to 80112.44]
  HPV 11 type antigen, Month 7: number analyzed (Participants) | 211 | 201 | 205 | 203
  HPV 11 type antigen, Month 7 | 276225.68 [243524.62 to 313317.91] | 250405.46 [217218.09 to 288663.30] | 260309.15 [223319.56 to 303425.52] | 187507.09 [162968.13 to 215740.99]
  HPV 11 type antigen, Month 12: number analyzed (Participants) | 210 | 209 | 205 | 205
  HPV 11 type antigen, Month 12 | 129019.87 [112127.85 to 148456.67] | 120984.83 [103575.25 to 141320.73] | 117640.77 [100745.01 to 137370.08] | 87423.54 [75807.40 to 100819.64]
  HPV 16 type antigen, Day 1: number analyzed (Participants) | 258 | 253 | 260 | 254
  HPV 16 type antigen, Day 1 | 684.26 [518.08 to 903.75] | 637.99 [490.56 to 829.73] | 690.99 [530.87 to 899.40] | 525.21 [416.24 to 662.71]
  HPV 16 type antigen, Month 2: number analyzed (Participants) | 231 | 227 | 230 | 229
  HPV 16 type antigen, Month 2 | 34918.40 [27711.11 to 44000.21] | 31250.65 [24952.39 to 39138.66] | 25605.94 [20018.80 to 32752.43] | 17397.59 [13647.75 to 22177.73]
  HPV 16 type antigen, Month 3: number analyzed (Participants) | 219 | 224 | 227 | 223
  HPV 16 type antigen, Month 3 | 252250.95 [217434.89 to 292641.82] | 217440.98 [184257.65 to 256600.37] | 201303.15 [171349.89 to 236492.48] | 158136.76 [134715.83 to 185629.53]
  HPV 16 type antigen, Month 6: number analyzed (Participants) | 219 | 214 | 217 | 208
  HPV 16 type antigen, Month 6 | 101518.07 [87448.85 to 117850.81] | 83015.52 [71509.49 to 96372.89] | 76558.80 [64740.19 to 90534.95] | 56636.27 [47641.12 to 67329.80]
  HPV 16 type antigen, Month 7: number analyzed (Participants) | 202 | 191 | 202 | 197
  HPV 16 type antigen, Month 7 | 297480.37 [254936.96 to 347123.34] | 272728.60 [231905.67 to 320737.69] | 294326.70 [252346.28 to 343290.99] | 154844.90 [131166.44 to 182797.86]
  HPV 16 type antigen, Month 12: number analyzed (Participants) | 205 | 202 | 203 | 201
  HPV 16 type antigen, Month 12 | 166953.66 [142318.06 to 195853.75] | 149269.66 [125174.31 to 178003.24] | 168097.78 [142244.20 to 198650.38] | 85986.11 [73074.57 to 101178.98]
  HPV 18 type antigen, Day 1: number analyzed (Participants) | 265 | 260 | 263 | 260
  HPV 18 type antigen, Day 1 | 1246.54 [1036.67 to 1498.89] | 1037.54 [885.47 to 1215.73] | 1111.98 [948.66 to 1303.41] | 952.51 [830.50 to 1092.44]
  HPV 18 type antigen, Month 2: number analyzed (Participants) | 236 | 233 | 231 | 233
  HPV 18 type antigen, Month 2 | 21700.85 [17733.79 to 26555.34] | 18029.88 [14988.53 to 21688.36] | 16571.70 [13555.92 to 20258.40] | 11081.57 [9094.95 to 13502.12]
  HPV 18 type antigen, Month 3: number analyzed (Participants) | 224 | 231 | 230 | 229
  HPV 18 type antigen, Month 3 | 137838.37 [118980.92 to 159684.56] | 127099.14 [108628.77 to 148710.05] | 123342.91 [106423.50 to 142952.21] | 79998.43 [68999.00 to 92751.33]
  HPV 18 type antigen, Month 6: number analyzed (Participants) | 226 | 221 | 219 | 212
  HPV 18 type antigen, Month 6 | 61676.34 [53576.84 to 71000.30] | 51216.03 [44364.44 to 59125.78] | 46904.59 [40385.36 to 54476.18] | 26774.11 [22940.11 to 31248.90]
  HPV 18 type antigen, Month 7: number analyzed (Participants) | 211 | 200 | 205 | 203
  HPV 18 type antigen, Month 7 | 181939.71 [157766.95 to 209816.17] | 172862.73 [148117.04 to 201742.65] | 183180.47 [156207.11 to 214811.50] | 86756.51 [73744.88 to 102063.92]
  HPV 18 type antigen, Month 12: number analyzed (Participants) | 210 | 208 | 205 | 205
  HPV 18 type antigen, Month 12 | 84949.48 [72424.07 to 99641.09] | 77008.45 [64999.61 to 91235.95] | 87334.91 [73919.46 to 103185.10] | 36658.81 [31077.43 to 43242.59]
  HPV 31 type antigen, Day 1: number analyzed (Participants) | 265 | 260 | 264 | 261
  HPV 31 type antigen, Day 1 | 2748.41 [2441.79 to 3093.53] | 2698.81 [2418.57 to 3011.52] | 2595.69 [2371.22 to 2841.42] | 2358.09 [2189.79 to 2539.33]
  HPV 31 type antigen, Month 2: number analyzed (Participants) | 236 | 234 | 234 | 234
  HPV 31 type antigen, Month 2 | 32102.49 [27409.98 to 37598.34] | 31733.68 [27111.16 to 37144.34] | 27652.57 [23288.94 to 32833.82] | 12606.73 [10568.61 to 15037.90]
  HPV 31 type antigen, Month 3: number analyzed (Participants) | 224 | 231 | 231 | 229
  HPV 31 type antigen, Month 3 | 161264.11 [142962.02 to 181909.25] | 146413.17 [128682.36 to 166587.07] | 133818.05 [117762.32 to 152062.83] | 89306.66 [79122.92 to 100801.13]
  HPV 31 type antigen, Month 6: number analyzed (Participants) | 226 | 221 | 220 | 212
  HPV 31 type antigen, Month 6 | 68516.79 [60395.61 to 77730.00] | 61717.39 [54357.98 to 70073.18] | 54672.61 [47682.67 to 62687.23] | 32131.34 [27928.72 to 36966.36]
  HPV 31 type antigen, Month 7: number analyzed (Participants) | 211 | 200 | 206 | 203
  HPV 31 type antigen, Month 7 | 241644.97 [215104.30 to 271460.37] | 221590.60 [192869.71 to 254588.41] | 230875.63 [202104.78 to 263742.19] | 104667.37 [90853.53 to 120581.53]
  HPV 31 type antigen, Month 12: number analyzed (Participants) | 205 | 207 | 204 | 204
  HPV 31 type antigen, Month 12 | 137744.87 [120414.00 to 157570.13] | 132414.54 [113520.94 to 154452.65] | 143396.41 [125201.11 to 164236.01] | 55178.34 [47206.87 to 64495.90]
  HPV 33 type antigen, Day 1: number analyzed (Participants) | 264 | 258 | 260 | 259
  HPV 33 type antigen, Day 1 | 624.29 [528.02 to 738.12] | 578.18 [489.56 to 682.84] | 566.26 [487.33 to 657.97] | 523.15 [456.49 to 599.54]
  HPV 33 type antigen, Month 2: number analyzed (Participants) | 235 | 231 | 230 | 233
  HPV 33 type antigen, Month 2 | 18225.37 [15231.33 to 21807.94] | 16873.64 [14013.68 to 20317.26] | 14523.05 [12060.26 to 17488.76] | 12110.80 [10065.98 to 14571.01]
  HPV 33 type antigen, Month 3: number analyzed (Participants) | 220 | 223 | 224 | 223
  HPV 33 type antigen, Month 3 | 124361.59 [108348.67 to 142741.07] | 113348.19 [96632.64 to 132955.20] | 105284.68 [90915.50 to 121924.92] | 87895.71 [76051.15 to 101585.00]
  HPV 33 type antigen, Month 6: number analyzed (Participants) | 215 | 212 | 201 | 204
  HPV 33 type antigen, Month 6 | 43736.52 [38187.42 to 50091.97] | 41162.19 [35659.00 to 47514.67] | 35892.14 [30909.82 to 41677.54] | 30563.15 [26208.11 to 35641.88]
  HPV 33 type antigen, Month 7: number analyzed (Participants) | 208 | 200 | 198 | 198
  HPV 33 type antigen, Month 7 | 154537.14 [133354.03 to 179085.17] | 146931.12 [125717.81 to 171723.90] | 150919.88 [128301.37 to 177525.85] | 96875.65 [84426.91 to 111159.96]
  HPV 33 type antigen, Month 12: number analyzed (Participants) | 209 | 207 | 202 | 203
  HPV 33 type antigen, Month 12 | 79450.21 [68289.18 to 92435.36] | 75043.46 [63377.35 to 88857.01] | 78826.94 [67275.95 to 92361.18] | 46210.95 [40274.75 to 53022.09]
  HPV 45 type antigen, Day 1 | 2431.92 [2233.39 to 2648.10] | 2408.58 [2235.09 to 2595.54] | 2315.53 [2182.69 to 2456.46] | 2217.15 [2109.75 to 2330.02]
  HPV 45 type antigen, Month 2: number analyzed (Participants) | 236 | 235 | 234 | 234
  HPV 45 type antigen, Month 2 | 17122.75 [14408.88 to 20347.76] | 17097.47 [14406.77 to 20290.70] | 14345.03 [12174.35 to 16902.74] | 6292.08 [5323.98 to 7436.22]
  HPV 45 type antigen, Month 3: number analyzed (Participants) | 224 | 232 | 231 | 229
  HPV 45 type antigen, Month 3 | 137598.43 [121615.96 to 155681.28] | 127933.76 [111246.84 to 147123.69] | 113479.94 [99528.64 to 129386.85] | 55337.26 [48187.68 to 63547.61]
  HPV 45 type antigen, Month 6: number analyzed (Participants) | 226 | 222 | 220 | 212
  HPV 45 type antigen, Month 6 | 45691.56 [40155.51 to 51990.83] | 41003.12 [35887.26 to 46848.26] | 34796.86 [30257.59 to 40017.12] | 16153.45 [13858.32 to 18828.69]
  HPV 45 type antigen, Month 7: number analyzed (Participants) | 211 | 201 | 206 | 203
  HPV 45 type antigen, Month 7 | 170959.55 [149389.05 to 195644.64] | 174740.31 [151200.15 to 201945.41] | 174014.45 [150322.39 to 201440.58] | 71768.92 [61224.65 to 84129.14]
  HPV 45 type antigen, Month 12: number analyzed (Participants) | 210 | 209 | 206 | 205
  HPV 45 type antigen, Month 12 | 78692.83 [68331.72 to 90624.98] | 80653.92 [68737.56 to 94636.11] | 82021.92 [70210.67 to 95820.12] | 29716.61 [25237.04 to 34991.31]
  HPV 52 type antigen, Day 1: number analyzed (Participants) | 265 | 260 | 264 | 260
  HPV 52 type antigen, Day 1 | 1641.65 [1464.30 to 1840.48] | 1720.51 [1525.62 to 1940.31] | 1611.71 [1461.90 to 1776.89] | 1549.58 [1410.22 to 1702.72]
  HPV 52 type antigen, Month 2: number analyzed (Participants) | 236 | 233 | 234 | 234
  HPV 52 type antigen, Month 2 | 75187.13 [66352.61 to 85197.91] | 83557.87 [73382.84 to 95143.74] | 73047.67 [63982.97 to 83396.59] | 25513.64 [21690.75 to 30010.30]
  HPV 52 type antigen, Month 3: number analyzed (Participants) | 224 | 231 | 231 | 228
  HPV 52 type antigen, Month 3 | 185490.54 [166270.48 to 206932.34] | 176024.77 [153898.90 to 201331.66] | 164122.51 [144482.99 to 186431.62] | 95239.18 [84388.59 to 107484.91]
  HPV 52 type antigen, Month 6: number analyzed (Participants) | 226 | 221 | 220 | 211
  HPV 52 type antigen, Month 6 | 75353.61 [66851.68 to 84936.78] | 77979.01 [68903.19 to 88250.29] | 65136.98 [56955.32 to 74493.93] | 32359.34 [28207.45 to 37122.36]
  HPV 52 type antigen, Month 7: number analyzed (Participants) | 211 | 200 | 206 | 201
  HPV 52 type antigen, Month 7 | 203994.24 [180491.88 to 230556.91] | 196454.98 [172561.35 to 223657.02] | 204005.75 [178367.04 to 233329.81] | 103497.80 [90571.68 to 118268.69]
  HPV 52 type antigen, Month 12: number analyzed (Participants) | 207 | 208 | 206 | 203
  HPV 52 type antigen, Month 12 | 123724.49 [107358.59 to 142585.25] | 131043.47 [113718.55 to 151007.84] | 129678.87 [113220.94 to 148529.14] | 54071.66 [46680.66 to 62632.89]
  HPV 58 type antigen, Day 1: number analyzed (Participants) | 265 | 261 | 263 | 261
  HPV 58 type antigen, Day 1 | 692.12 [578.03 to 828.72] | 615.45 [518.19 to 730.95] | 643.72 [548.71 to 755.18] | 571.59 [492.66 to 663.17]
  HPV 58 type antigen, Month 2: number analyzed (Participants) | 236 | 235 | 233 | 235
  HPV 58 type antigen, Month 2 | 35027.13 [29855.93 to 41094.00] | 33438.25 [28322.91 to 39477.45] | 30732.28 [26045.95 to 36261.80] | 13395.37 [11180.86 to 16048.50]
  HPV 58 type antigen, Month 3: number analyzed (Participants) | 224 | 232 | 230 | 229
  HPV 58 type antigen, Month 3 | 158592.29 [139984.81 to 179673.18] | 144355.15 [124064.76 to 167963.98] | 140028.57 [120462.67 to 162772.43] | 79942.78 [69460.78 to 92006.58]
  HPV 58 type antigen, Month 6: number analyzed (Participants) | 226 | 221 | 219 | 212
  HPV 58 type antigen, Month 6 | 70466.12 [61803.06 to 80343.50] | 66072.77 [57862.76 to 75447.68] | 57807.95 [49486.07 to 67529.30] | 33188.99 [28367.50 to 38829.98]
  HPV 58 type antigen, Month 7: number analyzed (Participants) | 210 | 199 | 205 | 202
  HPV 58 type antigen, Month 7 | 193735.34 [167223.71 to 224450.13] | 186513.90 [161169.95 to 215843.18] | 190767.16 [162753.08 to 223603.20] | 93456.26 [80147.35 to 108975.18]
  HPV 58 type antigen, Month 12: number analyzed (Participants) | 202 | 205 | 203 | 204
  HPV 58 type antigen, Month 12 | 114626.18 [98236.18 to 133750.73] | 110249.43 [93894.97 to 129452.48] | 115765.42 [99881.91 to 134174.76] | 51715.19 [44122.31 to 60614.71]

22. Secondary Outcome: Number of Participants With Seroconversion for Anti-HPV IgG Antibodies
Description: Seroconversion is defined as the appearance of antibodies [i.e., concentration greater than or equal to (>=) the lower limit of quantification (LLOQ) value] in the serum of participants seronegative [i.e, concentrations less than (<) the LLOQ value] before vaccination.
  The assessed antigens were: HPV 6, HPV 11, HPV 16, HPV 18, HPV 31, HPV 33, HPV 45, HPV 52 and HPV 58 type antigens.
  The LLOQ values specific to each antigen are as follows: HPV 6 type: LLOQ = 5100 AU/mL; HPV 11 type: LLOQ = 2480 AU/mL; HPV 16 type: LLOQ = 404 AU/mL; HPV 18 type: LLOQ = 1234 AU/mL; HPV 31 type: LLOQ = 3849 AU/mL; HPV 33 type: LLOQ = 617 AU/mL; HPV 45 type: LLOQ = 4079 AU/mL; HPV 52 type: LLOQ = 2352 AU/mL and HPV 58 type: LLOQ = 660 AU/mL.
Time Frame: At Month 2, Month 3, Month 6, Month 7 and Month 12
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 217 | 216 | 220 | 222
Participants
  HPV 6 type antigen, Month 2: number analyzed (Participants) | 199 | 200 | 209 | 219
  HPV 6 type antigen, Month 2 | 186 | 186 | 189 | 137
  HPV 6 type antigen, Month 3: number analyzed (Participants) | 190 | 201 | 207 | 213
  HPV 6 type antigen, Month 3 | 186 | 197 | 201 | 211
  HPV 6 type antigen, Month 6: number analyzed (Participants) | 190 | 193 | 198 | 198
  HPV 6 type antigen, Month 6 | 187 | 189 | 191 | 173
  HPV 6 type antigen, Month 7: number analyzed (Participants) | 181 | 177 | 184 | 191
  HPV 6 type antigen, Month 7 | 179 | 174 | 178 | 186
  HPV 6 type antigen, Month 12: number analyzed (Participants) | 168 | 174 | 178 | 184
  HPV 6 type antigen, Month 12 | 165 | 170 | 174 | 172
  HPV 11 type antigen, Month 2: number analyzed (Participants) | 200 | 196 | 195 | 211
  HPV 11 type antigen, Month 2 | 198 | 192 | 190 | 208
  HPV 11 type antigen, Month 3: number analyzed (Participants) | 194 | 195 | 196 | 207
  HPV 11 type antigen, Month 3 | 192 | 192 | 191 | 206
  HPV 11 type antigen, Month 6: number analyzed (Participants) | 191 | 187 | 188 | 190
  HPV 11 type antigen, Month 6 | 189 | 185 | 183 | 187
  HPV 11 type antigen, Month 7: number analyzed (Participants) | 184 | 174 | 174 | 184
  HPV 11 type antigen, Month 7 | 183 | 172 | 169 | 182
  HPV 11 type antigen, Month 12: number analyzed (Participants) | 179 | 177 | 174 | 185
  HPV 11 type antigen, Month 12 | 177 | 175 | 171 | 184
  HPV 16 type antigen, Month 2: number analyzed (Participants) | 170 | 164 | 171 | 178
  HPV 16 type antigen, Month 2 | 170 | 163 | 169 | 177
  HPV 16 type antigen, Month 3: number analyzed (Participants) | 166 | 164 | 172 | 173
  HPV 16 type antigen, Month 3 | 166 | 162 | 170 | 172
  HPV 16 type antigen, Month 6: number analyzed (Participants) | 161 | 155 | 166 | 164
  HPV 16 type antigen, Month 6 | 161 | 154 | 165 | 164
  HPV 16 type antigen, Month 7: number analyzed (Participants) | 156 | 145 | 152 | 157
  HPV 16 type antigen, Month 7 | 156 | 144 | 152 | 157
  HPV 16 type antigen, Month 12: number analyzed (Participants) | 155 | 148 | 152 | 160
  HPV 16 type antigen, Month 12 | 155 | 147 | 151 | 160
  HPV 18 type antigen, Month 2: number analyzed (Participants) | 190 | 192 | 188 | 197
  HPV 18 type antigen, Month 2 | 187 | 186 | 185 | 187
  HPV 18 type antigen, Month 3: number analyzed (Participants) | 185 | 192 | 188 | 193
  HPV 18 type antigen, Month 3 | 182 | 189 | 185 | 192
  HPV 18 type antigen, Month 6: number analyzed (Participants) | 182 | 184 | 181 | 179
  HPV 18 type antigen, Month 6 | 180 | 182 | 178 | 177
  HPV 18 type antigen, Month 7: number analyzed (Participants) | 175 | 170 | 167 | 172
  HPV 18 type antigen, Month 7 | 174 | 168 | 164 | 170
  HPV 18 type antigen, Month 12: number analyzed (Participants) | 172 | 176 | 166 | 174
  HPV 18 type antigen, Month 12 | 170 | 174 | 163 | 173
  HPV 31 type antigen, Month 2: number analyzed (Participants) | 203 | 197 | 196 | 208
  HPV 31 type antigen, Month 2 | 199 | 192 | 189 | 171
  HPV 31 type antigen, Month 3: number analyzed (Participants) | 196 | 196 | 196 | 203
  HPV 31 type antigen, Month 3 | 192 | 192 | 191 | 202
  HPV 31 type antigen, Month 6: number analyzed (Participants) | 195 | 188 | 189 | 187
  HPV 31 type antigen, Month 6 | 193 | 185 | 185 | 184
  HPV 31 type antigen, Month 7: number analyzed (Participants) | 187 | 173 | 174 | 180
  HPV 31 type antigen, Month 7 | 186 | 170 | 170 | 180
  HPV 31 type antigen, Month 12: number analyzed (Participants) | 180 | 178 | 173 | 179
  HPV 31 type antigen, Month 12 | 178 | 175 | 171 | 178
  HPV 33 type antigen, Month 2: number analyzed (Participants) | 170 | 173 | 171 | 181
  HPV 33 type antigen, Month 2 | 168 | 170 | 168 | 179
  HPV 33 type antigen, Month 3: number analyzed (Participants) | 161 | 169 | 169 | 173
  HPV 33 type antigen, Month 3 | 159 | 166 | 166 | 172
  HPV 33 type antigen, Month 6: number analyzed (Participants) | 155 | 160 | 155 | 159
  HPV 33 type antigen, Month 6 | 153 | 158 | 152 | 157
  HPV 33 type antigen, Month 7: number analyzed (Participants) | 155 | 159 | 151 | 157
  HPV 33 type antigen, Month 7 | 154 | 157 | 148 | 156
  HPV 33 type antigen, Month 12: number analyzed (Participants) | 155 | 161 | 153 | 161
  HPV 33 type antigen, Month 12 | 153 | 159 | 151 | 161
  HPV 45 type antigen, Month 2 | 190 | 190 | 191 | 122
  HPV 45 type antigen, Month 3: number analyzed (Participants) | 206 | 213 | 218 | 217
  HPV 45 type antigen, Month 3 | 203 | 206 | 213 | 212
  HPV 45 type antigen, Month 6: number analyzed (Participants) | 207 | 203 | 208 | 200
  HPV 45 type antigen, Month 6 | 204 | 200 | 203 | 179
  HPV 45 type antigen, Month 7: number analyzed (Participants) | 194 | 188 | 194 | 192
  HPV 45 type antigen, Month 7 | 192 | 185 | 189 | 188
  HPV 45 type antigen, Month 12: number analyzed (Participants) | 194 | 193 | 194 | 194
  HPV 45 type antigen, Month 12 | 191 | 190 | 190 | 184
  HPV 52 type antigen, Month 2: number analyzed (Participants) | 205 | 200 | 200 | 201
  HPV 52 type antigen, Month 2 | 202 | 198 | 197 | 194
  HPV 52 type antigen, Month 3: number analyzed (Participants) | 198 | 200 | 199 | 196
  HPV 52 type antigen, Month 3 | 196 | 195 | 195 | 194
  HPV 52 type antigen, Month 6: number analyzed (Participants) | 197 | 191 | 190 | 185
  HPV 52 type antigen, Month 6 | 195 | 190 | 187 | 182
  HPV 52 type antigen, Month 7: number analyzed (Participants) | 188 | 177 | 177 | 175
  HPV 52 type antigen, Month 7 | 186 | 176 | 175 | 173
  HPV 52 type antigen, Month 12: number analyzed (Participants) | 183 | 181 | 177 | 177
  HPV 52 type antigen, Month 12 | 180 | 180 | 174 | 175
  HPV 58 type antigen, Month 2: number analyzed (Participants) | 182 | 183 | 173 | 186
  HPV 58 type antigen, Month 2 | 180 | 180 | 170 | 186
  HPV 58 type antigen, Month 3: number analyzed (Participants) | 175 | 184 | 174 | 181
  HPV 58 type antigen, Month 3 | 173 | 181 | 170 | 180
  HPV 58 type antigen, Month 6: number analyzed (Participants) | 174 | 176 | 167 | 169
  HPV 58 type antigen, Month 6 | 172 | 174 | 163 | 168
  HPV 58 type antigen, Month 7: number analyzed (Participants) | 166 | 164 | 155 | 162
  HPV 58 type antigen, Month 7 | 165 | 162 | 152 | 161
  HPV 58 type antigen, Month 12: number analyzed (Participants) | 158 | 166 | 153 | 165
  HPV 58 type antigen, Month 12 | 156 | 164 | 151 | 164

23. Secondary Outcome: Anti-HPV Neutralizing Titers
Description: Anti-HPV neutralizing titers were determined by pseudovirion-based neutralization (PBNA) assay and expressed as geometric mean titers (GMTs). The assessed antigens were: HPV 6, HPV 11, HPV 16, HPV 18, HPV 31, HPV 33, HPV 45, HPV 52 and HPV 58 type antigens.
Time Frame: At Day 1, Month 3 and Month 7
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 266 | 261 | 264 | 261
Titers
  HPV 6 type antigen, Day 1 | 328.72 [265.51 to 406.99] | 280.37 [232.07 to 338.73] | 242.72 [206.00 to 286.00] | 230.40 [196.29 to 270.43]
  HPV 6 type antigen, Month 3: number analyzed (Participants) | 223 | 229 | 227 | 226
  HPV 6 type antigen, Month 3 | 45690.44 [39581.97 to 52741.61] | 41126.63 [35026.80 to 48288.74] | 39346.74 [33229.37 to 46590.30] | 21637.85 [18354.48 to 25508.56]
  HPV 6 type antigen, Month 7: number analyzed (Participants) | 149 | 140 | 147 | 141
  HPV 6 type antigen, Month 7 | 82061.27 [70437.95 to 95602.62] | 75228.75 [61603.93 to 91866.94] | 71805.19 [57989.96 to 88911.69] | 33651.69 [27317.93 to 41453.96]
  HPV 11 type antigen, Day 1 | 225.65 [193.18 to 263.58] | 210.97 [183.33 to 242.77] | 204.12 [178.72 to 233.13] | 189.59 [168.38 to 213.47]
  HPV 11 type antigen, Month 3: number analyzed (Participants) | 224 | 231 | 228 | 228
  HPV 11 type antigen, Month 3 | 13233.27 [11647.45 to 15035.00] | 12081.23 [10600.08 to 13769.35] | 10838.85 [9463.76 to 12413.73] | 11547.59 [10251.71 to 13007.27]
  HPV 11 type antigen, Month 7: number analyzed (Participants) | 149 | 140 | 147 | 142
  HPV 11 type antigen, Month 7 | 17321.54 [14965.94 to 20047.91] | 16793.17 [14214.38 to 19839.80] | 16315.93 [13807.32 to 19280.31] | 12607.96 [10724.69 to 14821.94]
  HPV 16 type antigen, Day 1 | 361.27 [291.97 to 447.02] | 325.48 [270.30 to 391.92] | 356.83 [294.43 to 432.46] | 277.19 [236.97 to 324.24]
  HPV 16 type antigen, Month 3: number analyzed (Participants) | 224 | 232 | 231 | 229
  HPV 16 type antigen, Month 3 | 35416.74 [29603.66 to 42371.29] | 31018.79 [26065.77 to 36912.98] | 29774.15 [24560.51 to 36094.53] | 21870.13 [18225.32 to 26243.85]
  HPV 16 type antigen, Month 7: number analyzed (Participants) | 149 | 140 | 147 | 142
  HPV 16 type antigen, Month 7 | 83674.41 [68253.56 to 102579.36] | 75779.10 [59852.62 to 95943.55] | 81101.64 [64972.49 to 101234.78] | 37820.19 [29988.35 to 47697.42]
  HPV 18 type antigen, Day 1 | 73.24 [61.47 to 87.27] | 63.14 [54.42 to 73.25] | 64.18 [55.86 to 73.73] | 57.05 [50.67 to 64.22]
  HPV 18 type antigen, Month 3: number analyzed (Participants) | 225 | 232 | 230 | 229
  HPV 18 type antigen, Month 3 | 3994.46 [3295.05 to 4842.33] | 3610.97 [3001.43 to 4344.30] | 3528.45 [2908.77 to 4280.15] | 1705.98 [1394.09 to 2087.65]
  HPV 18 type antigen, Month 7: number analyzed (Participants) | 149 | 140 | 147 | 142
  HPV 18 type antigen, Month 7 | 9236.06 [7400.65 to 11526.67] | 9539.94 [7507.03 to 12123.35] | 9756.59 [7610.84 to 12507.29] | 3518.33 [2745.04 to 4509.45]
  HPV 31 type antigen, Day 1 | 86.49 [72.60 to 103.02] | 85.98 [71.95 to 102.75] | 86.03 [73.71 to 100.41] | 76.01 [66.25 to 87.22]
  HPV 31 type antigen, Month 3: number analyzed (Participants) | 225 | 232 | 231 | 229
  HPV 31 type antigen, Month 3 | 22472.04 [19266.57 to 26210.81] | 21241.61 [17729.34 to 25449.67] | 18317.84 [15540.80 to 21591.12] | 9156.79 [7772.33 to 10787.86]
  HPV 31 type antigen, Month 7: number analyzed (Participants) | 149 | 140 | 147 | 142
  HPV 31 type antigen, Month 7 | 69730.78 [56719.94 to 85726.14] | 64413.46 [49797.87 to 83318.69] | 59252.25 [46942.33 to 74790.26] | 17581.92 [14014.44 to 22057.53]
  HPV 33 type antigen, Day 1 | 207.88 [185.90 to 232.47] | 216.99 [191.26 to 246.17] | 200.17 [181.73 to 220.49] | 186.32 [172.16 to 201.64]
  HPV 33 type antigen, Month 3: number analyzed (Participants) | 225 | 232 | 230 | 229
  HPV 33 type antigen, Month 3 | 17034.78 [14730.51 to 19699.52] | 15199.08 [12954.60 to 17832.44] | 12923.25 [10949.50 to 15252.79] | 9132.50 [7752.49 to 10758.18]
  HPV 33 type antigen, Month 7: number analyzed (Participants) | 149 | 140 | 147 | 142
  HPV 33 type antigen, Month 7 | 33246.87 [27979.03 to 39506.53] | 30752.43 [25717.48 to 36773.13] | 27855.80 [22482.02 to 34514.06] | 18696.71 [15656.33 to 22327.51]
  HPV 45 type antigen, Day 1 | 55.65 [48.99 to 63.21] | 61.43 [53.20 to 70.94] | 53.80 [48.31 to 59.93] | 49.89 [45.89 to 54.25]
  HPV 45 type antigen, Month 3: number analyzed (Participants) | 225 | 232 | 230 | 229
  HPV 45 type antigen, Month 3 | 13822.73 [11844.34 to 16131.59] | 13197.57 [11085.72 to 15711.73] | 11113.74 [9429.52 to 13098.77] | 3488.90 [2963.94 to 4106.83]
  HPV 45 type antigen, Month 7: number analyzed (Participants) | 149 | 139 | 146 | 142
  HPV 45 type antigen, Month 7 | 25204.55 [20693.56 to 30698.90] | 24537.36 [20030.78 to 30057.86] | 22748.14 [18260.65 to 28338.42] | 7853.20 [6210.60 to 9930.24]
  HPV 52 type antigen, Day 1 | 78.63 [68.76 to 89.92] | 85.37 [73.69 to 98.89] | 75.58 [67.66 to 84.43] | 72.37 [64.86 to 80.75]
  HPV 52 type antigen, Month 3: number analyzed (Participants) | 225 | 232 | 231 | 229
  HPV 52 type antigen, Month 3 | 18288.04 [16184.95 to 20664.41] | 15548.20 [13427.71 to 18003.57] | 14606.62 [12634.89 to 16886.04] | 7903.98 [6883.36 to 9075.93]
  HPV 52 type antigen, Month 7: number analyzed (Participants) | 149 | 140 | 147 | 142
  HPV 52 type antigen, Month 7 | 21604.03 [18522.86 to 25197.74] | 20617.17 [17543.87 to 24228.84] | 20285.76 [17088.28 to 24081.54] | 10904.65 [9006.10 to 13203.43]
  HPV 58 type antigen, Day 1 | 87.31 [72.70 to 104.85] | 87.15 [72.02 to 105.46] | 82.06 [69.30 to 97.16] | 73.81 [63.25 to 86.13]
  HPV 58 type antigen, Month 3: number analyzed (Participants) | 225 | 232 | 231 | 229
  HPV 58 type antigen, Month 3 | 31623.27 [27319.75 to 36604.69] | 27936.10 [23519.92 to 33181.47] | 27246.89 [22979.23 to 32307.15] | 11650.18 [9904.82 to 13703.09]
  HPV 58 type antigen, Month 7: number analyzed (Participants) | 149 | 140 | 147 | 142
  HPV 58 type antigen, Month 7 | 51354.94 [42792.24 to 61631.03] | 46896.70 [38584.84 to 56999.07] | 46983.15 [37929.98 to 58197.15] | 22245.13 [18114.56 to 27317.58]

24. Secondary Outcome: Anti-HPV Neutralizing Titers in a Subset of Participants
Description: Anti-HPV neutralizing titers were determined by PBNA assay and expressed as GMTs. The assessed antigens were: HPV 6, HPV 11, HPV 16, HPV 18, HPV 31, HPV 33, HPV 45, HPV 52 and HPV 58 type antigens.
Time Frame: At Month 2
Population: Analysis was performed on a subset of participants from Per Protocol Set (PPS) for immunogenicity with post-vaccination immunogenicity results available for the specified analysis at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 92 | 91 | 89 | 88
Titers
  HPV 6 type antigen: number analyzed (Participants) | 84 | 82 | 82 | 80
  HPV 6 type antigen | 13438.35 [9145.74 to 19745.74] | 11275.45 [7643.73 to 16632.69] | 6658.75 [4614.67 to 9608.24] | 3364.11 [2041.48 to 5543.64]
  HPV 11 type antigen | 2592.37 [1870.39 to 3593.02] | 2441.65 [1755.07 to 3396.81] | 1531.82 [1119.26 to 2096.46] | 2912.25 [2156.54 to 3932.76]
  HPV 16 type antigen | 5888.86 [3547.05 to 9776.79] | 4711.97 [2939.99 to 7551.96] | 2947.73 [1742.01 to 4987.98] | 2987.06 [1757.29 to 5077.45]
  HPV 18 type antigen | 603.31 [365.97 to 994.56] | 447.98 [286.20 to 701.20] | 379.32 [237.94 to 604.69] | 259.14 [161.99 to 414.56]
  HPV 31 type antigen | 4005.68 [2737.23 to 5861.95] | 3612.79 [2463.24 to 5298.82] | 2193.35 [1620.34 to 2969.00] | 1183.70 [775.15 to 1807.59]
  HPV 33 type antigen | 1830.91 [1260.56 to 2659.31] | 1782.19 [1234.63 to 2572.59] | 1097.86 [810.20 to 1487.66] | 1182.00 [818.69 to 1706.55]
  HPV 45 type antigen | 1382.24 [973.72 to 1962.14] | 1657.88 [1178.35 to 2332.56] | 1119.04 [824.21 to 1519.32] | 369.17 [267.20 to 510.05]
  HPV 52 type antigen | 9664.68 [7775.37 to 12013.06] | 9081.81 [7013.61 to 11759.89] | 8379.90 [6544.29 to 10730.38] | 4052.45 [3070.88 to 5347.77]
  HPV 58 type antigen | 5169.27 [3769.39 to 7089.05] | 5519.36 [3960.66 to 7691.47] | 3848.83 [2823.14 to 5247.19] | 1569.91 [1070.81 to 2301.63]

25. Secondary Outcome: Number of Participants With Seroconversion for Anti-HPV Neutralizing Antibodies
Description: Seroconversion is defined as the appearance of antibodies (i.e., titer >=LLOQ value) in the serum of participants seronegative (i.e, titer <LLOQ value) before vaccination.
  The assessed antigens were: HPV 6, HPV 11, HPV 16, HPV 18, HPV 31, HPV 33, HPV 45, HPV 52 and HPV 58 type antigens.
  The LLOQ values specific to each antigen are as follows: HPV 6 type: LLOQ = 269 titers; HPV 11 type: LLOQ = 279 titers; HPV 16 type: LLOQ = 339 titers; HPV 18 type: LLOQ = 84 titers; HPV 31 type: LLOQ = 96 titers; HPV 33 type: LLOQ = 323 titers; HPV 45 type: LLOQ = 76 titers; HPV 52 type: LLOQ = 104 titers and HPV 58 type: LLOQ = 95 titers.
Time Frame: At Month 3 and Month 7
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 208 | 211 | 216 | 217
Participants
  HPV 6 type antigen, Month 3: number analyzed (Participants) | 173 | 182 | 186 | 194
  HPV 6 type antigen, Month 3 | 172 | 179 | 181 | 192
  HPV 6 type antigen, Month 7: number analyzed (Participants) | 112 | 111 | 120 | 120
  HPV 6 type antigen, Month 7 | 112 | 109 | 116 | 119
  HPV 11 type antigen, Month 3: number analyzed (Participants) | 199 | 200 | 203 | 208
  HPV 11 type antigen, Month 3 | 195 | 196 | 198 | 206
  HPV 11 type antigen, Month 7: number analyzed (Participants) | 132 | 121 | 132 | 129
  HPV 11 type antigen, Month 7 | 130 | 118 | 128 | 127
  HPV 16 type antigen, Month 3: number analyzed (Participants) | 189 | 188 | 191 | 199
  HPV 16 type antigen, Month 3 | 187 | 185 | 187 | 196
  HPV 16 type antigen, Month 7: number analyzed (Participants) | 125 | 111 | 115 | 123
  HPV 16 type antigen, Month 7 | 124 | 109 | 114 | 121
  HPV 18 type antigen, Month 3: number analyzed (Participants) | 195 | 204 | 198 | 203
  HPV 18 type antigen, Month 3 | 192 | 199 | 193 | 195
  HPV 18 type antigen, Month 7: number analyzed (Participants) | 131 | 122 | 123 | 123
  HPV 18 type antigen, Month 7 | 129 | 119 | 120 | 120
  HPV 31 type antigen, Month 3: number analyzed (Participants) | 190 | 188 | 187 | 192
  HPV 31 type antigen, Month 3 | 189 | 184 | 186 | 192
  HPV 31 type antigen, Month 7: number analyzed (Participants) | 120 | 109 | 116 | 118
  HPV 31 type antigen, Month 7 | 120 | 107 | 116 | 118
  HPV 33 type antigen, Month 3 | 204 | 206 | 210 | 215
  HPV 33 type antigen, Month 7: number analyzed (Participants) | 139 | 123 | 140 | 132
  HPV 33 type antigen, Month 7 | 136 | 121 | 135 | 131
  HPV 45 type antigen, Month 3: number analyzed (Participants) | 187 | 188 | 192 | 188
  HPV 45 type antigen, Month 3 | 185 | 184 | 189 | 186
  HPV 45 type antigen, Month 7: number analyzed (Participants) | 124 | 113 | 122 | 117
  HPV 45 type antigen, Month 7 | 122 | 111 | 119 | 116
  HPV 52 type antigen, Month 3: number analyzed (Participants) | 188 | 191 | 193 | 194
  HPV 52 type antigen, Month 3 | 186 | 188 | 189 | 193
  HPV 52 type antigen, Month 7: number analyzed (Participants) | 121 | 112 | 119 | 118
  HPV 52 type antigen, Month 7 | 120 | 111 | 118 | 116
  HPV 58 type antigen, Month 3: number analyzed (Participants) | 195 | 192 | 195 | 195
  HPV 58 type antigen, Month 3 | 193 | 188 | 190 | 193
  HPV 58 type antigen, Month 7: number analyzed (Participants) | 128 | 116 | 121 | 118
  HPV 58 type antigen, Month 7 | 126 | 114 | 118 | 116

26. Secondary Outcome: Correlation Between Anti-HPV IgG Antibody Concentration and Anti-HPV Neutralizing Antibody Titers
Description: The Pearson coefficient of correlation between anti-HPV IgG antibody concentration and anti-HPV neutralizing antibody titers was calculated for each study group and for each antigen. The Pearson correlation was computed by the log10-transformation of specific antibody concentrations.
Time Frame: At Day 1, Month 2, Month 3 and Month 7
Population: Analysis was performed on a subset of participants from Per Protocol Set for analysis of immunogenicity, which included participants with both concentration and titer values available for the specified analysis at the specified time points. Participants with values below the LLOQ or above ULOQ in either assay were excluded from the analysis.
Measure: Number; unit: Correlation coefficient
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
Number analyzed (Participants) | 211 | 223 | 213 | 225
Correlation coefficient
  HPV 6 type antigen, Day 1: number analyzed (Participants) | 42 | 37 | 28 | 21
  HPV 6 type antigen, Day 1 | 0.850 | 0.818 | 0.756 | 0.830
  HPV 6 type antigen, Month 2: number analyzed (Participants) | 61 | 66 | 70 | 48
  HPV 6 type antigen, Month 2 | 0.824 | 0.851 | 0.766 | 0.786
  HPV 6 type antigen, Month 3: number analyzed (Participants) | 175 | 185 | 190 | 203
  HPV 6 type antigen, Month 3 | 0.813 | 0.790 | 0.789 | 0.867
  HPV 6 type antigen, Month 7: number analyzed (Participants) | 95 | 81 | 89 | 118
  HPV 6 type antigen, Month 7 | 0.820 | 0.810 | 0.786 | 0.892
  HPV 11 type antigen, Day 1: number analyzed (Participants) | 30 | 30 | 32 | 26
  HPV 11 type antigen, Day 1 | 0.907 | 0.921 | 0.951 | 0.932
  HPV 11 type antigen, Month 2: number analyzed (Participants) | 73 | 72 | 73 | 75
  HPV 11 type antigen, Month 2 | 0.840 | 0.831 | 0.807 | 0.820
  HPV 11 type antigen, Month 3: number analyzed (Participants) | 173 | 176 | 182 | 187
  HPV 11 type antigen, Month 3 | 0.806 | 0.808 | 0.820 | 0.856
  HPV 11 type antigen, Month 7: number analyzed (Participants) | 91 | 79 | 86 | 104
  HPV 11 type antigen, Month 7 | 0.659 | 0.839 | 0.787 | 0.820
  HPV 16 type antigen, Day 1: number analyzed (Participants) | 49 | 51 | 54 | 40
  HPV 16 type antigen, Day 1 | 0.934 | 0.927 | 0.918 | 0.951
  HPV 16 type antigen, Month 2: number analyzed (Participants) | 80 | 79 | 70 | 73
  HPV 16 type antigen, Month 2 | 0.965 | 0.951 | 0.880 | 0.958
  HPV 16 type antigen, Month 3 | 0.871 | 0.862 | 0.827 | 0.904
  HPV 16 type antigen, Month 7: number analyzed (Participants) | 143 | 133 | 138 | 135
  HPV 16 type antigen, Month 7 | 0.866 | 0.893 | 0.894 | 0.894
  HPV 18 type antigen, Day 1: number analyzed (Participants) | 38 | 31 | 39 | 30
  HPV 18 type antigen, Day 1 | 0.903 | 0.863 | 0.896 | 0.920
  HPV 18 type antigen, Month 2: number analyzed (Participants) | 61 | 65 | 64 | 54
  HPV 18 type antigen, Month 2 | 0.885 | 0.885 | 0.811 | 0.866
  HPV 18 type antigen, Month 3: number analyzed (Participants) | 203 | 212 | 203 | 213
  HPV 18 type antigen, Month 3 | 0.881 | 0.880 | 0.860 | 0.884
  HPV 18 type antigen, Month 7: number analyzed (Participants) | 130 | 127 | 117 | 133
  HPV 18 type antigen, Month 7 | 0.899 | 0.871 | 0.881 | 0.905
  HPV 31 type antigen, Day 1: number analyzed (Participants) | 34 | 38 | 42 | 25
  HPV 31 type antigen, Day 1 | 0.751 | 0.811 | 0.708 | 0.344
  HPV 31 type antigen, Month 2: number analyzed (Participants) | 83 | 84 | 83 | 77
  HPV 31 type antigen, Month 2 | 0.768 | 0.820 | 0.824 | 0.745
  HPV 31 type antigen, Month 3: number analyzed (Participants) | 194 | 207 | 208 | 218
  HPV 31 type antigen, Month 3 | 0.800 | 0.800 | 0.798 | 0.845
  HPV 31 type antigen, Month 7: number analyzed (Participants) | 107 | 96 | 101 | 127
  HPV 31 type antigen, Month 7 | 0.814 | 0.824 | 0.806 | 0.842
  HPV 33 type antigen, Day 1: number analyzed (Participants) | 22 | 23 | 20 | 15
  HPV 33 type antigen, Day 1 | 0.664 | 0.843 | 0.831 | 0.886
  HPV 33 type antigen, Month 2: number analyzed (Participants) | 65 | 69 | 68 | 63
  HPV 33 type antigen, Month 2 | 0.794 | 0.790 | 0.672 | 0.711
  HPV 33 type antigen, Month 3: number analyzed (Participants) | 184 | 188 | 194 | 203
  HPV 33 type antigen, Month 3 | 0.811 | 0.767 | 0.783 | 0.859
  HPV 33 type antigen, Month 7: number analyzed (Participants) | 80 | 78 | 77 | 114
  HPV 33 type antigen, Month 7 | 0.649 | 0.807 | 0.789 | 0.768
  HPV 45 type antigen, Day 1: number analyzed (Participants) | 19 | 23 | 18 | 14
  HPV 45 type antigen, Day 1 | 0.721 | 0.885 | 0.692 | 0.557
  HPV 45 type antigen, Month 2: number analyzed (Participants) | 78 | 77 | 73 | 57
  HPV 45 type antigen, Month 2 | 0.834 | 0.859 | 0.740 | 0.805
  HPV 45 type antigen, Month 3: number analyzed (Participants) | 192 | 193 | 199 | 220
  HPV 45 type antigen, Month 3 | 0.846 | 0.863 | 0.799 | 0.882
  HPV 45 type antigen, Month 7: number analyzed (Participants) | 86 | 74 | 87 | 127
  HPV 45 type antigen, Month 7 | 0.869 | 0.870 | 0.737 | 0.882
  HPV 52 type antigen, Day 1: number analyzed (Participants) | 31 | 37 | 39 | 28
  HPV 52 type antigen, Day 1 | 0.809 | 0.790 | 0.847 | 0.804
  HPV 52 type antigen, Month 2: number analyzed (Participants) | 77 | 76 | 78 | 78
  HPV 52 type antigen, Month 2 | 0.748 | 0.832 | 0.606 | 0.767
  HPV 52 type antigen, Month 3: number analyzed (Participants) | 149 | 151 | 172 | 203
  HPV 52 type antigen, Month 3 | 0.797 | 0.821 | 0.754 | 0.861
  HPV 52 type antigen, Month 7: number analyzed (Participants) | 77 | 70 | 67 | 113
  HPV 52 type antigen, Month 7 | 0.777 | 0.834 | 0.829 | 0.831
  HPV 58 type antigen, Day 1: number analyzed (Participants) | 40 | 35 | 38 | 31
  HPV 58 type antigen, Day 1 | 0.632 | 0.816 | 0.791 | 0.831
  HPV 58 type antigen, Month 2: number analyzed (Participants) | 79 | 77 | 85 | 80
  HPV 58 type antigen, Month 2 | 0.666 | 0.733 | 0.666 | 0.803
  HPV 58 type antigen, Month 3: number analyzed (Participants) | 169 | 172 | 171 | 210
  HPV 58 type antigen, Month 3 | 0.831 | 0.721 | 0.789 | 0.852
  HPV 58 type antigen, Month 7: number analyzed (Participants) | 63 | 69 | 67 | 121
  HPV 58 type antigen, Month 7 | 0.851 | 0.860 | 0.825 | 0.851

ADVERSE EVENTS:
Time Frame: Solicited AEs: during the 7-day follow-up period after any vaccination. Unsolicited AEs: during the 28-day follow-up period after any vaccination. All-cause mortality, SAEs and pIMDs: from first vaccination (Day 1) up to study end (Month 12).
Description: All events presented in the All-cause mortality, Serious Adverse Events and Other (not including Serious) Adverse Events modules are reported for the Exposed Set population during the specified time frames.
Arm/Group | HPV9 High Group | HPV9 Med Group | HPV9 Low Group | Gar9 Group
All-Cause Mortality (participants affected / at risk) | 0/270 | 0/270 | 0/269 | 0/270
Serious Adverse Events (participants affected / at risk) | 1/270 | 4/270 | 2/269 | 7/270
Other Adverse Events (participants affected / at risk) | 260/270 | 265/270 | 262/269 | 254/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPV9 High Group (N=270) | HPV9 Med Group (N=270) | HPV9 Low Group (N=269) | Gar9 Group (N=270)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bartholin's abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Personality disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal septal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPV9 High Group (N=270) | HPV9 Med Group (N=270) | HPV9 Low Group (N=269) | Gar9 Group (N=270)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 5 (6) | 3 (6) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (4)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polycystic ovarian syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (4) | 5 (5) | 9 (10)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 5 (5) | 1 (1) | 3 (3)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 6 (6) | 2 (2) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (14) | 5 (5) | 15 (21) | 7 (7)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (2) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (4) | 1 (1)
Administration site erythema (General disorders) | 126 (211) | 131 (217) | 139 (224) | 89 (130)
Administration site pain (General disorders) | 255 (636) | 262 (656) | 256 (654) | 235 (528)
Administration site swelling (General disorders) | 113 (188) | 99 (161) | 106 (183) | 59 (80)
Asthenia (General disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Fatigue (General disorders) | 213 (458) | 205 (402) | 192 (373) | 192 (379)
Induration (General disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (2)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (5)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Injection site granuloma (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Injection site induration (General disorders) | 4 (5) | 0 (0) | 1 (1) | 3 (5)
Injection site mass (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site pain (General disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (2)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 34 (38) | 37 (37) | 25 (31) | 33 (37)
Swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site bruising (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaccination site induration (General disorders) | 1 (1) | 3 (4) | 4 (4) | 2 (4)
Vaccination site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 6 (6) | 5 (5) | 2 (2) | 7 (7)
Cystitis (Infections and infestations) | 1 (1) | 9 (9) | 1 (1) | 3 (3)
Enterovirus infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (11) | 5 (6) | 10 (11) | 6 (6)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (3) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 4 (4) | 1 (3) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 4 (4) | 6 (6) | 5 (5)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 17 (17) | 11 (11) | 11 (15) | 15 (16)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood prolactin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Human papilloma virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 (75) | 44 (60) | 47 (65) | 45 (56)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4) | 5 (5)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 137 (228) | 133 (231) | 126 (213) | 118 (178)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 4 (4)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 194 (384) | 180 (319) | 187 (354) | 179 (337)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5) | 3 (3)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thoracic radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 13 (13) | 11 (14) | 11 (17) | 9 (9)
Menstruation delayed (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3) | 4 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other symptoms/illnesses or reactions (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT05496231/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT05496231/SAP_001.pdf